## NCT02819310

## STUDY PROTOCOL

# An Open Label Study of Chronic Use of BLI400 Laxative in Constipated Adults

**DOCUMENT DATE: 04/13/2016** 


Braintree Laboratories, Inc. Protocol Number BL1400-303

## An Open Label Study of Chronic Use of BLI400 Laxative in Constipated Adults

#### Braintree Protocol BLI400-303

Version Dated 4-13-2016

**SPONSOR** 

Braintree Laboratories, Inc. 60 Columbian St. West P.O. Box 850929
Braintree, MA 02185
PH: 781-843-2301

Mark Cleveland

Sr. Vice President, R&D/RA

Braintree Laboratories, Inc.

Principal Investigator

Michael P. DeMicco, MD, FACG, ABAM

Anahiem Clinical Trials, LLC

4/14/16

Date

Date

| 1. | INTRO | ODUCTION | 5 |
|---|---|---|---|
| 2. | STUD | Y OBJECTIVE | 10 |
| 3. | | Y PLAN | |
| | | rudy Design | |
| | | UMBER OF SUBJECTS | |
| | | URATION OF STUDY | |
| | | ΓUDY TREATMENTS | |
| | 3.5. St | UBJECT SELECTION | 12 |
| | <i>3.5.1</i> . | Inclusion Criteria | 12 |
| | <i>3.5.2.</i> | Exclusion Criteria | 13 |
| 4. | STUD | Y PROCEDURES | 14 |
| | 4.1. V | ISIT 1 (DAY 0) | 14 |
| | <i>4.1.1</i> . | Informed Consent | |
| | <i>4.1.2.</i> | Enrollment and Allocation of Subject Number | 15 |
| | <i>4.1.3</i> . | Study Drug | |
| | | REATMENT PERIOD | |
| | 4.2.1. | Treatment Day 1 | |
| | 4.2.2. | Visit 2 (Month 2) +/- 4 days | |
| | 4.2.3. | Visit 3 (Month 4) +/- 4 days | |
| | <i>4.2.4. 4.2.5.</i> | Visit 4 (Month 6) +/- 4 days<br>Visit 5 (Month 9) +/- 4 days | |
| | 4.2.5.<br>4.2.6. | Visit 6 (Month 12 or Early Term) +/- 4 days | |
| | 4.2.7. | Follow-up Telephone Call (Day 374) +/- 4 days | |
| | | ABULATED STUDY PROCEDURES | |
| | | REGNANCY | |
| | 4.5. Co | ONCOMITANT MEDICATIONS | 20 |
| 5. | ADVE | RSE EVENTS | 21 |
| | 5.1. A | DVERSE EVENT DEFINITION AND REPORTING | 21 |
| 6. | SERIC | OUS ADVERSE EVENTS REPORTING | 23 |
| 7. | | TUTIONAL REVIEW BOARD AND INFORMED CONSENT | |
| <b>8.</b> | | AGEMENT OF INTERCURRENT EVENTS | |
| | | ODIFICATION OF PROTOCOL | |
| _ | | | |
| 9. | | ANALYSIS | |
| | | AMPLE SIZE | |
| | | ARAMETERS TO BE ANALYZED | |
| | | LANNED ANALYSES | |
| | 9.3.1. | Demographic and Baseline Characteristics | |
| | 9.3.2.<br>9.3.3. | Safety Analyses Efficacy Analyses (Patient Reported Outcomes) | |
| | 7.J.J. | Lijikuky Anutyses (1 utent Keporteu Outkomes) | •••••• <u>4</u> / |

#### Braintree Laboratories, Inc. Protocol Number BLI400-303

#### Confidential

| 9.4. S | STUDY POPULATIONS | 27 |
|---------|-----------------------------------------------|----|
| | Intention-to-Treat (ITT) Population | |
| | Modified Intention-to-Treat (mITT) Population | |
| 9.4.2. | Per-Protocol Population | 28 |
| 10. DR | UG INVENTORY AND DISPOSITION | 28 |
| 11. ST | UDY MONITORING | 28 |
| 12. DO | CUMENTS AND NOTIFICATIONS | 28 |
| 12.1. I | NFORMED CONSENT | 28 |
| 12.2. I | NSTITUTIONAL REVIEW BOARD | 28 |
| 12.3. A | AMENDMENTS TO THE PROTOCOL | 29 |
| 12.4. I | Data Records | 29 |
| 13. PU | BLICATION AND AGREEMENT | 29 |
| 14. INV | VESTIGATORS AGREEMENT | 30 |
| 15. RE | FERENCES | 31 |
| 16. AP | PENDIX A | 32 |
| API | PENDIX B | 35 |

BLI400 (NDA 211281)

Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

#### CLINICAL PROTOCOL SUMMARY SHEET

#### **STUDY TITLE:**

An Open Label Study of Chronic Use of BLI400 Laxative in Constipated Adults

**PROTOCOL:** BLI400-303

**VERSION DATE:** 4-13-2016

**IND NUMBER:** 118,906

#### **OBJECTIVE:**

To evaluate the safety of chronic use of BLI400 Laxative in constipated adults.

#### STUDY DESIGN:

This is an open-label, multi-center study in constipated outpatients.

#### **SUBJECTS:**

Approximately 300 male or female adult subjects with a history of constipation will be enrolled in this study (including approximately 100 elderly subjects).

#### **STUDY MEDICATIONS:**

BLI400 Laxative (21 grams of Lactitol Monohydrate, NF)

#### **DURATION OF TREATMENT**

Subjects will take BLI400 laxative daily for 12 months (52 weeks). Participation in this study will last for approximately 54 weeks, including the 14 day follow up telephone call.

#### PRIMARY ENDPOINT

Safety will be analyzed through the use of adverse event and ECG data, and the comparison of chemistry, hematology, and urinalysis values as measured at baseline and at specific time points throughout the study.

#### 1. INTRODUCTION

The present approaches to the treatment of chronic idiopathic constipation (CIC) are limited and for some patients there are significant drawbacks that have not been resolved. It would be desirable to provide a source of relief for constipation that would permit dosing adjustments to optimize efficacy and safety and that would be pleasant to consume to improve patient compliance. The treatment should not have the safety issues associated with oral phosphate laxatives, have an acceptable safety profile, and be effective in numerous types of constipation.

Braintree Laboratories, Inc. is investigating the use of a new chemical composition, BLI400 (Lactitol Monohydrate NF Powder for Reconstitution) as a treatment for adult constipation. Ample published literature with lactitol provides significant preclinical and clinical studies which support the safe and effective use of this GRAS-listed compound.

These reports indicate that the BLI400 lactitol composition has promise as a candidate for further development for the treatment of constipation, as reviewed herein.

BLI400 is a member of the pharmaceutical class of osmotic laxatives; specifically it is a non-absorbed, colonically metabolized sugar alcohol (polyol). Studies reviewed here indicate it provides relief from the symptoms of constipation by rapidly inducing a patient-controlled bowel movement. While lactitol appears to be minimally, if at all, absorbed in the small intestine, colonic microbes split lactitol into D-galactose and D-sorbitol, which are fermentable to organic acids including lactic, formic, propionic, butyric and acetic acids (as reviewed in Patil et al, 1987). The osmotic properties of the small organic molecules consistently point to their pharmacodynamic effects as dependent on water retention with the stool. Thus, BLI400 is a pro-drug of an essentially non-absorbed osmotic laxative. Lactitol is generally considered to be pharmacologically inert and is often referred to as a "prebiotic" with no specific receptor targets for its laxative action.

#### Rationale for Performing Research with the Investigational Product

Lactitol monohydrate, at a daily dose of 21 grams per day appears to be a safe and effective treatment for constipation, but it has not been studied and proven in clinical

Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

trials in the US. Lactitol appears to be a "prebiotic", a substrate for colonic bacteria which convert it into osmotically active small molecules. Extensive published and non-published literature supports its safety and efficacy, but a Phase III clinical trial is required for its registration in the US. It is envisaged there will be one, multi-site, controlled study in patients with documented constipation and that the design will be similar to other studies that have led to the approval of laxatives, such as those for MiraLAX, NDA 22-015 and consistent with FDA's recommendations for study endpoints in CIC trials.

#### Physical, Chemical, and Pharmaceutical Properties and Formulation

Lactitol is a simple monosaccharide sugar alcohol, a synthetic derivative of the milk sugar lactose that was discovered in the 1920s. It is a dry, free flowing powder, readily soluble in aqueous solutions. As shown by the structure diagrams, it is an analog of the disaccharide lactulose.

Lactitol

Lactulose

Table 1-1
Components of a Typical Single Dose of BLI400

| Component | Amount (g)* |
|--------------------------|-------------|
| Lactitol monohydrate, NF | 21 |

The product will be provided in multi-dose bottles with a measuring cap to deliver 10.5 grams of BLI400.

**Nonclinical Studies:** Extensive nonclinical studies have been performed with lactitol as support for its registration and marketing in countries outside the US and are reviewed in detail in the BLI400 Investigators' Brochure. The studies have covered basic pharmacology, genotoxicity and mutagenicity, acute and chronic studies including carcinogenicity and reproductive toxicity. These studies were carried out in mice, rats, dogs and rabbits.

**Pharmacology:** Lactitol is not degraded by the galactosidase enzymes of the small intestine However, colonic microflora degrade lactitol extensively in rats so that lactitol elevated the proportions of acetic acid and lowered proportions of butyric acid in the hindgut of rats. The osmotic effects of these organic acids appear to provide the pharmacodynamic basis for lactitol's laxative action. Increased output of moist feces was seen in all animals species studied in a dose-related manner. The highest doses tested caused frank diarrhea in some studies.

**Metabolic Effects:** In some studies, total serum cholesterol and triglycerides were reduced equally in rats fed diets containing 7% sorbitol or lactitol. By acidifying fecal contents, lactitol lowered ammonia levels in animal models of hepatic encephalopathy, perhaps as a result of production of the poorly absorbed ammonium ion that follows lowering the cecal pH. Rats fed a diet containing 5% of lactitol for two weeks displayed a significant increase of calcium absorption.

Toxicology Studies: Only weak edema ensued after lactitol application to intact skin, but erythema and edema emerged when it was applied to abraded skin. Rodents treated with lactitol had loose, frequent stools and cecal enlargement. This was often accompanied by decreased weight gain and increased water consumption. Clinical chemistry changes included changes in electrolyte levels, decreased cholesterol and alkaline phosphatase. Perhaps as compensation for the electrolyte changes that probably followed the diarrhea, adrenal weight and hypertrophy of the zona fasciculata were seen in the highest dose groups. Renal tubular degeneration with nephrocalcinosis was occasionally seen and may follow the increased calcium absorption. Lactitol was not considered positive for mutagenicity or chromosomal damage studied in standard in vitro and in vivo assays. Life-long carcinogenicity studies have indicated that Leydig cell dysplasia occurred in

rats at high lactitol doses, but this was not seen in mice dosed for 24 months or dogs dosed for 12 months. This species-specific effect in some rat strains was not considered significant to humans, since ordinary milk sugar, lactose, produces a similar effect in rodents.

Clinical Pharmacology and Safety: Since lactitol is extensively degraded to organic acids in the colon, it is little surprise that there are no published studies on its level in blood after administration. Some have estimated that only 0.6% of an oral dose of lactitol is excreted in urine. Similar to what is found in animals, lactitol is extensively metabolized in the human colon, making available a significant proportion of the metabolites for colonic absorption. Unlike in animals, lactitol does not seem to stimulate calcium absorption in humans, although in one study when 15 g of lactitol was administered along with calcium in solution to fasting volunteers, calcium absorption was diminished. Administering lactitol increases fecal Bifidobacteria levels, while other bacteria (fecal anaerobes, aerobes, Enterobacteriaceae or lactobacilli) were unaffected. After the ingestion of 25 g lactitol, xylitol, or glucose by eight healthy male volunteers the rise in plasma glucose was significantly greater 30 and 60 minutes after ingestion of glucose while no rise in plasma glucose followed ingestion of lactitol.

The investigation of the use of a mixture of lactitol for the treatment of constipation has been extensively studied, but the information is only available in published form. From these observations, it appears that lactitol's adverse events are limited largely to the gastrointestinal system. Symptoms such as nausea, cramps, abdominal pain, flatulence and vomiting may be expected and could lead to withdrawal from the study if not controlled. Their incidence and severity may be ameliorated in some patients by dose-adjustment. Changes in hematology, clinical chemistry or urinalysis may be seen, and their clinical significance will be assessed during the development of lactitol. In one study plasma potassium was elevated with lactitol, but the values stayed within the normal range.

Clinical Efficacy: Lactitol has been marketed since at least 1985 outside the US in Europe and other regions (where it is known as Lactitol Ex-Lax® or Importal®, for example) as a syrup or powder for the treatment of constipation in adults, including the elderly and children. As a result a substantial body of evidence has accumulated on its

use in treating constipation, as evidenced by more than 19 publications since 1988, including two recent review articles (Maydeo, 2010; Faruqui and Joshi, 2012).

A minimal effective dose of 0.25 g/kg has been suggested, and most studies have found that a starting dose of 20 g of lactitol is effective and produces minimal side effects. Some studies that have allowed the subjects to make dosage increases to achieve relief of constipation symptoms and dose reductions to minimize side effects have indicated that this strategy can optimize therapy.

Maydeo (2010) presented a systematic review of six published randomized, non-randomized and open trials comparing the safety and efficacy of lactitol to those of lactulose. Overall, lactitol was comparable to lactulose in efficacy measures (normal stool consistency and number of bowel movement per week). Patients found lactitol to be more acceptable and were more compliant with it largely due to its superior palatability (73.2 % vs. 26.8 %). Lactitol was significantly better than lactulose in the frequency of adverse events  $(31.2 \pm 0.8 \% \text{ vs. } 62.1 \pm 1.1 \%, p=0.0019)$ . The physicians' assessment favored lactitol as compared to lactulose (61.91% vs. 47.83%). The following table is adapted from Maydeo's summary of the reviewed trials.

| Parameter Evaluated | Lactitol | Lactulose |
|--------------------------------------|------------------|---------------|
| Patient's acceptance | 73.2% | 26.8% |
| Consistency of stool (normal/soft) | $80.5 \pm 4.5\%$ | 75.0± 8.0% |
| Bowel movement/week | $5.9 \pm 0.2$ | $5.6 \pm 0.6$ |
| Incidence of side-effects | $31.2 \pm 0.8$ | 62.1 ±1.1% |
| Global efficacy judged by physicians | 61.9% | 47.8% |


#### 2. STUDY OBJECTIVE

To evaluate the safety of chronic use of BLI400 laxative in constipated adults.

#### 3. STUDY PLAN

#### 3.1. Study Design

This is an open-label, multi-center study in which constipated subjects will receive BLI400 for 12 months.

#### 3.2. Number of Subjects

Approximately 300 constipated subjects will be enrolled into this study, including approximately 100 elderly subjects ( $\geq$  65 years of age at Visit 1).

#### 3.3. Duration of Study

Qualifying subjects will receive BLI400 at Visit 1 and will begin a 12-month Treatment Period. Subjects will return for clinic visits at the end of Months 2, 4, 6, 9 and 12. A follow up call will take place 2 weeks after the end of treatment. A completed subject is defined as a subject that completes the Visit 6 (Month 12) visit.

#### 3.4. Study Treatments

#### **BLI400 Laxative**

BLI400 laxative will be provided polyethylene bottles containing sufficient study medication for 30 days of dosing. The bottles will be equipped with a cap that can be used to measure 10.5 grams of BLI400. Each bottle will also have a clinical label containing a caution statement, study code, study sponsor and subject number. Subjects will be instructed to mix the contents of 2 capfuls (approximately 21 g) in 4 - 8 oz of juice or other beverage, and take once daily preferably in the morning. Subjects that develop persistent diarrhea or loose stools will be allowed to adjust their dose down to 10.5g (1 capful) per day.

#### **Rescue Bisacodyl**

Subjects will be dispensed bisacodyl at each study visit (previously dispensed bisacodyl may be redispensed if needed, although this is not encouraged). Subjects will be instructed to take 5 - 10 mg (1 - 2 tablets) of bisacodyl if they are experiencing severe discomfort due to their constipation, or have not had a BM in 4 days. No more than 6 tablets (30mg) of bisacodyl should be taken in a week.

If a subject does not have a bowel movement within 24 hours of taking a bisacodyl dose, a second dose should be taken. If after the second bisacodyl dose the subject does not have a BM within 24 hours, the subject should contact the site. The investigator should then consider having the subject return for an evaluation and/or discontinuing the subject from the study.

All study medication is required to remain at room temperature 20°-25°C (68°-77°F); excursions permitted between 15°-30°C (59°-86°F).


#### 3.5. Subject Selection

#### 3.5.1. Inclusion Criteria

Subjects will be admitted to the study if they are:

- 1. Male or female subjects at least 18 years of age
- 2. Constipated, defined by the following adapted ROME II definition (Drossman et al, 2000):
  - A. Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for at least 12 weeks (which need not be consecutive) in the preceding 12 months:
    - a. Straining during > 25% of defecations
    - b. Lumpy or hard stools in > 25% of defecations
    - c. Sensation of incomplete evacuation for > 25% of defecations
- 3. If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, sterilized, abstinent, or vasectomized spouse)
- 4. Negative urine pregnancy test at screening, if applicable
- 5. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Braintree Laboratories, Inc. Protocol Number BLI400-303


#### 3.5.2. Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

- 1. Report loose (mushy) or water stools in the absence of laxative use for more than 25% of BMs during the 12 weeks before Visit 1
- 2. Meet the Rome II criteria for Irritable Bowel Syndrome: reports abdominal discomfort or pain that has two or more of the following three features for at least 12 weeks, which need not be consecutive, in the 12 months before Visit 1:
  - Relieved with defecation
  - Onset associated with a change in frequency of stool
  - Onset associated with a change in form (appearance of stool)
- 3. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
- 4. Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
- 5. Subjects with hypothyroidism that is being treated and for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of Visit 1
- 6. Subjects taking laxatives, enemas or prokinetic agents that refuse to discontinue these treatments from Visit 1 until after completion of Visit 6
- 7. Subjects who are pregnant or lactating, or intend to become pregnant during the study
- 8. Subjects of childbearing potential who refuse a pregnancy test
- 9. Subjects who are allergic to any BLI400 component (lactitol)
- 10. Subjects taking narcotic analysis or other medications known to cause constipation.
- 11. Subjects with clinically significant cardiac abnormalities identified at the Visit 1 ECG
- 12. Subjects with clinically significant laboratory abnormalities, deemed as a potential safety issue by the Investigator, may be discontinued at the Investigator's discretion.
- 13. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
- 14. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
- 15. Subjects with an active history of drug or alcohol abuse
- 16. Subjects have been hospitalized for a psychiatric condition or have made a suicide attempt during the 2 years before Visit 1
- 17. Subjects who withdraw consent at any time prior to completion of Visit 1 procedures

Braintree Laboratories, Inc. Protocol Number BLI400-303


#### 4. STUDY PROCEDURES

Study procedures are described as follows and depicted graphically in Section 4.3, below. Acceptable deviations from the visit schedule are indicated. These variations must not be cumulative; i.e. visits should always be scheduled in relationship to Visit 1 (Day 0).

## 4.1. Visit 1 (Day 0)

At the screening visit, the following procedures will be undertaken:

- Subject is fully informed about the study and gives written agreement to study participation in the form of a signed informed consent form (refer to Section 4.1.1)
- Assess eligibility (refer to inclusion/exclusion criteria)
- Review of medications
- Medical history including history of constipation (ROME criteria See Inclusion #2)
- Physical examination
- Vital signs, including assessment of orthostatic hypotension (while seated and after standing for a minimum of 2 minutes) including height and bodyweight, pulse and temperature
- A 12-lead ECG will be performed by qualified, trained site personnel. ECG output must be reviewed by a physician investigator. Any clinically significant cardiac abnormalities identified on the ECG should disqualify a subject. Data from the ECG will be collected in the eCRF.
- Urine pregnancy test (if applicable)
- Blood and urine samples will be collected for testing at a central laboratory, as shown below.

<u>Chemistry:</u> alkaline phosphatase, ALT, anion gap, AST, bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatine kinase, creatinine, eGFR, GGT, HCG, inorganic phosphate, magnesium, osmolality, potassium, sodium, uric acid. CK-MB will be tested in samples where the CK value is greater than 2.5 times the upper normal limit.

<u>Hematology:</u> hematocrit, hemoglobin, platelets count, red blood cell count, white blood cell count (and differentials)

<u>Urinalysis:</u> including electrolytes (sodium, potassium, magnesium, calcium), microscopic analysis, urine osmolality

Subjects with clinically significant laboratory abnormalities, deemed as a potential safety issue by the Investigator, may be discontinued at the Investigator's discretion.

If the subject is eligible for the study, assign a subject number.

- Subjects will complete the Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL, refer to Appendix A) and the Patient Assessment of Constipation Symptom questionnaire (PAC-SYM, refer to Appendix B)
- Dispense 2 bottles of BLI400
- Dispense rescue bisacodyl. Subjects will be allowed to take 5 10mg of bisacodyl if they
  are experiencing severe discomfort due to their constipation, or have not had a BM in 4
  days.
- Instruct subject to maintain their normal dietary habits during study participation
- Schedule the next study visit to occur after 60 days

Subjects that are ineligible due to prohibited medication use (Exclusion Criterion 10) may be washed out for a period of 14 days. No additional procedures should be performed on these subjects. After the washout period, subjects may be enrolled and all Visit 1 procedures should be repeated (with the exception of obtaining informed consent).

#### 4.1.1. **Informed Consent**

Following the informed consent process, study subjects will sign a current IRB approved consent form. No study procedures may be performed prior to the subject providing informed consent. The subject's original signed and personally dated Informed Consent Form (together with any subsequent IRB approved amended versions) must be retained by the Investigator in the subject's file. A copy of the original signed and dated Informed Consent Form must be given to the subject.

#### 4.1.2. Enrollment and Allocation of Subject Number

Subjects will be enrolled into the study only when they have given their written, informed consent to participate.

Subjects enrolled at the screening visit will be assigned a subject number by site personnel.

This number will consist of:

- The 3-digit Site Number;
- The 3-digit subject identifier number (this number is a sequentially allocated number). Each site will begin with 001 for the first subject screened, 002 for the second and so on. For example, the third subject screened at Site 15 will become Subject Number 15-003. After a subject completes all screening procedures and eligibility has been confirmed, site personnel will assign a subject number.

#### 4.1.3. Study Drug

After it has been confirmed that all eligibility criteria have been met, site personnel will utilize the IWRS to assign a drug kit number to the subject.

Site personnel must only dispense the drug kit that has been assigned by the IWRS. Dispensing of incorrect kits is considered a protocol violation.

Subjects will be provided instructions on how to take the study medication and rescue medication. Two bottles will be dispensed per subject. The study drug bottles will be weighed for drug accountability purposes. Subjects will be instructed to return all bottles at each follow up visit.

#### 4.2. Treatment Period

#### 4.2.1. Treatment Day 1

Starting on the morning of Treatment Day 1 (the day after Visit 1), subjects will measure 2 capfuls of study medication and ingest it mixed in a beverage of their choice. Subject will take a daily dose of 2 capfuls until they return for Visit 2. Subjects that develop persistent diarrhea or loose stools should contact their study center. These subjects will be allowed to adjust their dose down to 10.5g (1 capful) per day.

#### 4.2.2. Visit 2 (Month 2) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 2 (Day 60). Vital signs (see section 4.1 for details) and ECGs will be recorded. Study personnel will weigh returned bottles and count rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Subjects will be dispensed 2 new bottles of study medication. Subjects will be instructed to return all bottles and bisacodyl at the next follow up visit.

Braintree Laboratories, Inc. Protocol Number BLI400-303


#### 4.2.3. Visit 3 (Month 4) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 3 (Day 120). Vital signs (See section 4.1 for details) will be recorded. Study personnel will weigh returned bottles and count rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Subjects will be dispensed 2 new bottles of study medication. Subjects will be instructed to return all bottles and bisacodyl at the next follow up visit.

#### 4.2.4. Visit 4 (Month 6) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 4 (Day 180). Vital signs (See section 4.1 for details) will be recorded. Study personnel will review returned bottles and rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Subjects will be dispensed 3 new bottles of study medication. Subjects will be instructed to return all bottles and bisacodyl at the next follow up visit.

#### 4.2.5. Visit 5 (Month 9) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 5 (Day 270). Vital signs (See section 4.1 for details) will be recorded. Study personnel will review returned bottles and rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Three new bottles of study medication will be dispensed at this visit. Subjects will be instructed to return all bottles and bisacodyl at Visit 6.

#### 4.2.6. Visit 6 (Month 12 or Early Term) +/- 4 days

Subjects will return at Day 360 for their final clinic visit. Vital signs (see section 4.1 for details) and ECGs will be recorded. A physical examination will be performed. Study

personnel will weigh returned bottles and count bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Clinically significant laboratory abnormalities present at Visit 6 should be followed until resolved or are considered stable.

## 4.2.7. Follow-up Telephone Call (Day 374) +/- 4 days

At Day 374, approximately 2 weeks after the last study visit or early term visit, site personnel will contact subjects by telephone to query if any new adverse events have occurred and if any adverse events ongoing at Visit 6 have resolved. Subjects will also be asked about the status of their concomitant medications.

Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

## 4.3. Tabulated Study Procedures

The following graphically depicts the flow of study procedures at each visit.

| Procedures | Visit 1<br>Day 0 | Visit 2<br>Month 2<br>+/- 4 days | Visit 3<br>Month 4<br>+/- 4 days | Visit 4<br>Month 6<br>+/- 4 days | Visit 5<br>Month 9<br>+/- 4 days | Visit 6<br>Month 12/<br>ET<br>+/- 4 days | <b>☎</b> Day 374 +/- 4 days |
|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | 17- <b>4</b> uuys | |
| Inclusion/Exclusion Criteria Review | X | | | | | | |
| Medical History | X | | | | | | |
| Physical Examination | X | | | | | X | |
| Vital Signs <sup>1</sup> | X | X | X | X | X | X | |
| Electrocardiogram | X | X | | | | X | |
| Review of Concomitant Medication | X | X | X | X | X | X | X |
| Urine Pregnancy Test (if applicable) <sup>2</sup> | X | | | | | | |
| Enroll Eligible Subjects | X | | | | | | |
| Subject to Complete PAC-QOL, PAC-SYM | X | X | X | X | X | X | |
| Blood Sample for Chemistry Testing | X | X | X | X | X | X | |
| Blood Sample for Hematology Testing | X | X | X | X | X | X | |
| Urine Sample for Urinalysis | X | X | X | X | X | X | |
| Blood Sample for Serum Pregnancy Testing | | | | X | | X | |
| Dispense Study Drug and Rescue Bisacodyl | X | X | X | X | X | | |
| Study Drug and Rescue Bisacodyl Accountability | | X | X | X | X | X | |
| Assess Safety | | X | X | X | X | X | X |

blood pressure and pulse while seated and after standing for 2 minutes, temperature, weight and height (@Visit 1

<sup>&</sup>lt;sup>2</sup>only) refer to Section 4.4

#### 4.4. Pregnancy

Subjects who are female and of childbearing potential must have a urine pregnancy test done at screening. A positive result will rule out the participation of the subject in the study. Serum pregnancy tests will be performed at Visits 4 (Month 6) and 6 (Month 12). If a subject becomes pregnant during the study, the subject must be removed from the study and followed until one month after the end of the pregnancy.

Female study subjects must be surgically sterilized or using oral contraceptives, depot contraceptives, double-barrier method, intrauterine device, or testifies that she is monogamous with a vasectomized partner. Subjects practicing abstinence must agree to use an acceptable form of birth control should they become sexually active during the study.

Women with a history of bilateral tubal ligation are not considered of childbearing potential and are not required to have a urine pregnancy test at screening.

Oral contraceptives, hormone implants, and injections are only considered effective if started at least 1 month before the study.

Menopausal status is defined when menses have been absent for 12 months in a woman of appropriate age (usually 45 to 55 years) who has no other suspected or identified cause of amenorrhea.

#### 4.5. Concomitant Medications

The use of concomitant medication will be recorded from 7 days prior to Visit 1 until the end of the study at the telephone contact on Day 374. Subjects enrolled in this study will not be permitted to take any laxatives (other than the sponsor supplied rescue bisacodyl), whether prescription or over-the-counter, from Visit 1 until after completion of Visit 6. Any restricted laxative use during the study may result in termination of subject's participation. Subjects may not initiate treatment with any constipating medication.

#### 5. **ADVERSE EVENTS**

#### 5.1. Adverse Event Definition and Reporting

An Adverse Event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product.

Adverse event collection will coincide with the subject providing informed consent to participate in the study and will conclude with the end of study participation at Day 374 Follow-up Call. Diarrhea should be reported as an adverse event if a subject has more than 3 watery stools per day. Subjects with clinically significant laboratory results at Visit 6 which are classified by the Investigator as adverse events should return for a repeat blood draw. Subjects will be instructed to report promptly adverse events to the Investigator. The Investigator will record date/time of report, date/time of onset, description of the adverse event, severity of adverse event, action(s) taken regarding treatment of the event, action(s) taken regarding study participation, duration of adverse event, and the Investigator's assessment of relationship of adverse event to study treatment.

The Investigator should assess the severity of each adverse event using the following categories:

| Grade | Severity | Description |
|---|---|---|
| 1 | Mild | Barely noticeable, does not influence functioning |
| | MIIId | Causing no limitations of usual activities |
| 2 | Moderate | Makes participant uncomfortable, influences functioning |
| | Moderate | Causing some limitations of usual activities |
| 3 | | Severe discomfort, treatment needed |
| | Severe | Severe and undesirable, causing inability to carry out usual |
| | | activities |
| 4 | Life | Immediate risk of death |
| | threatening | Life threatening or disabling |
| 5 | Fatal | Causes death of the participant |

The Investigator should assess the relationship to study drug for each adverse event using the following categories:

| Categories of Attribution: | Description |
|---|---|
| UNRELATED | There is <i>no</i> evidence of any causal relationship. |
| POSSIBLE | There is <i>some</i> evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, the influence of <i>other factors may have contributed</i> to the event (e.g., the patient's clinical condition, other concomitant events). |
| PROBABLE | There <i>is evidence</i> to suggest a causal relationship, and the influence of other factors is <i>unlikely</i> . |
| DEFINITE | There is <i>clear</i> evidence to suggest a causal relationship, and other possible contributing factors can be <i>ruled out</i> . |

In published Phase 3 studies, adverse events associated with BLI400 administered at doses required for effective treatment of constipation included flatulence, nausea, vomiting, abdominal cramping or pain and bloating. These adverse reactions were transient and subsided rapidly upon dose adjustment or cessation.

#### 6. SERIOUS ADVERSE EVENTS REPORTING

A Serious Adverse Event (SAE) is any untoward medical occurrence that results in at least one of the following outcomes:

- Results in death
- Is life-threatening
- Requires inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly/birth defect
- Requires medical or surgical intervention to prevent permanent impairment or damage

SAE collection will coincide with the subject providing informed consent to participate in the study and will conclude 30 days after a subject's last dose of study medication. Should a serious and/or unexpected adverse event occur, the Investigator must notify Braintree Laboratories immediately. The Investigator will make a decision regarding continuing the subject's study participation, and may request input from Braintree Laboratories. The Investigator will be responsible for recommending or providing the subject with appropriate medical therapy. All subjects experiencing serious adverse events will be followed until satisfactory resolution occurs. Braintree Laboratories must be kept apprised of all follow-ups relative to serious adverse events. In addition, Investigators must comply with the SAE reporting requirements of the Institutional Review Board with oversight of the study.

Any serious and/or unexpected adverse events that occur during the study will be reported to Braintree Laboratories as follows:

Contact Telephone Numbers:

During Business hours 781-843-2301

(M-F, 8:30 am - 5:00 pm EDT)

After hours or weekends 781-964-9051

Braintree Laboratories and its medical monitor will review the report and determine whether an FDA Form 3500A will also be completed and sent to FDA.

#### 7. INSTITUTIONAL REVIEW BOARD AND INFORMED CONSENT

Institutional Review Board (IRB) review and approval of the study protocol and Informed Consent Form will be obtained prior to initiation of the study. Amendments to the study protocol and consent form generated during the course of the study will also require IRB approval.

#### 8. MANAGEMENT OF INTERCURRENT EVENTS

#### 8.1. Modification of Protocol

Neither an Investigator nor Braintree Laboratories will modify the protocol without first obtaining the concurrence of the other and the IRB. Investigators that continually violate the protocol or commit a serious violation may be subject to termination from the study. The study may be halted if at any time an Investigator or Braintree Laboratories deems the incidence or severity of adverse events to be unacceptable.

#### 8.2. Subjects Discontinued from the Study

Subjects may be dropped from the study for any of the following reasons:

- 1) Subject took prohibited medications during the Treatment Period
- 2) An adverse event requiring discontinuation (including failure to tolerate study medication).
- 3) The Investigator decides that the subject should be dropped from the study (e.g. serious adverse event, protocol violation, non-compliance).
- 4) The subject decides to withdraw from the study. Subjects are free to withdraw their consent and discontinue participation in the study at any time.

Braintree Laboratories should be contacted if possible prior to discontinuation of any subject. If a subject is discontinued from the study, Braintree Laboratories must be notified with an explanation for all discontinuances.

#### 9. DATA ANALYSIS

## 9.1. Sample Size

Consistent with ICH E1A Guideline for Industry, the Extent of Population Exposure to Assess Clinical Safety: for Drugs Intended for Long-term Treatment of Non-Life-Threatening Conditions (March 1995), 300 subjects will be treated with BLI400 for 12 months. This will allow for detection of adverse events that may increase in frequency or severity over time.

#### 9.2. Parameters to be Analyzed

The primary objective of this study is to investigate the safety of BLI400 used chronically for 12 months in subjects with constipation. Safety will be analyzed using ECG, vital signs, chemistry, hematology and urinalysis and adverse event data. Treatment emergent adverse event rates will be descriptively presented by preferred term, severity, and relationship to treatment.

#### 9.3. Planned Analyses

#### 9.3.1. Demographic and Baseline Characteristics

Baseline demographic characteristics will be tabulated with N, mean, standard deviation, and range of values where appropriate

- Age
- Gender
- Race/ethnicity
- Constipation History

#### 9.3.2. Safety Analyses

Analysis of safety will be performed using the modified Intent to Treat population (see Section 9.4).

#### Adverse Events

Adverse Events will be coded using the MedDRA classification to provide a preferred term and primary system organ class for each event. Proportions of subjects with adverse events will be presented for the overall study population, and each demographic subgroup (age, gender and race). Tables of AEs will be presented by system organ class and preferred term, and include overall totals for AEs within each system organ class. Counting will be done by subject and not by event. A table of counts and percentages will also be made of those subjects with SAEs or AEs which led to withdrawal from the study.

Treatment-emergent AEs are defined as adverse events that had an onset day and time on or after the day and time of the first dose of study drug until the Day 374 Follow-up Call. Adverse Events having missing onset dates will be considered as treatment emergent.

The difference in adverse event rates between study periods will be tested by Chi-Square or Fisher's exact test with 95% confidence intervals.

#### Laboratory Parameters

Summary statistics (i.e., mean, minimum, maximum, standard deviation, and number of subjects) will be presented for each laboratory parameter at each visit. Laboratory data will be summarized for the overall population and the elderly and non-elderly subgroups. When calculating the summary statistics only, the last observation within a visit window will be used if there are multiple observations. Changes from baseline (Visit 1) will be presented in a similar format. An additional listing will be provided of those subjects who have clinically significant laboratory values. The data will also be presented as shift tables and clinically significant abnormalities will be examined.

Results of laboratory tests for the change from baseline (Visit 1) and group differences will be tested using ANOVA.

#### Vital Signs

Summary statistics (i.e., mean, minimum, maximum, standard deviation, and number of subjects) will be presented for each vital sign at each visit and compared to the values obtained at Visit 1. When calculating the summary statistics only, the last observation within a visit window will be used if there are multiple observations. The data will also be presented as shift tables and clinically significant abnormalities will be examined.

ECG variables will be tabulated and presented for data collected at each visit. Data will be tabulated and summarized with descriptive statistics (N, mean, SD, CV%, SEM, minimum, and maximum) for each of the ECG variables. The differences in ECG variables between Visit 1 (Baseline), Visit 2 and Visit 6 will be tested using ANOVA.

#### 9.3.3. Efficacy Analyses (Patient Reported Outcomes)

Subject constipation symptoms and quality of life indicators will be analyzed using data from the subject-completed PAC-SYM and PAC-QOL instruments. Change from baseline to each visit time point will be presented for each collected measure and will be tested using ANOVA. Data for each measure and time point will also be presented categorically by severity and tested using Chi-Square or Fisher's exact test.

#### 9.4. Study Populations

The following populations have been defined for data analyses.

#### 9.4.1.Intention-to-Treat (ITT) Population

This population includes all enrolled subjects that were dispensed study medication.

#### 9.4.1. Modified Intention-to-Treat (mITT) Population

This population consists of all enrolled subjects that took at least one dose of study medication. This population will be utilized for all safety analyses.

#### 9.4.2. **Per-Protocol Population**

The per-protocol (PP) population will consist of all subjects in the mITT population who have not violated study entry criteria and have not deviated significantly from the protocol during the course of the study. Any analyses from this population will be considered as supportive to the ITT and mITT analyses. Reasons for exclusion from the PP population will be defined in the clinical study report.

#### 10. DRUG INVENTORY AND DISPOSITION

At the conclusion of the study, all drug materials will be accounted for. Federal law requires that, at the conclusion of the study, all drug materials must be returned to the study sponsor or destroyed according to local regulations.

#### 11. STUDY MONITORING

A Braintree Laboratories Study Monitor or qualified designee will visit the study center prior to the commencement of the study and periodically during the course of the study in accordance with federal guidelines governing the sponsorship of studies.

#### 12. DOCUMENTS AND NOTIFICATIONS

#### 12.1. Informed Consent

Written informed consent will be obtained from the subjects by the Investigator and will be kept on file at the study center. Documentation of the consent process should be noted in the study source documents.

#### 12.2. Institutional Review Board

Peer review and approval of the protocol by an appropriate Institutional Review Board is required prior to commencement of enrollment. Amendments to the approved protocol must also be submitted to the Institutional Review Board and approved prior to their implementation.

#### 12.3. Amendments to the Protocol

The Investigator and Braintree Laboratories will discuss any amendments to the study protocol. If an agreement is reached regarding the need for the amendment, it will be produced in writing by Braintree Laboratories and will be made a formal part of the protocol only after approval by an Institutional Review Board.

#### 12.4. Data Records

Site personnel will be required to enter study data into electronic case report forms (eCRFs) provided by Braintree Laboratories. Subject medical records will be reviewed to verify study data points, including potential adverse events, and to ensure correctness and consistency with the CRF entries. The Investigator should retain copies of paper and electronic data, patient consent/assent forms, and other study documents for a period of two years following the date of approval of a New Drug Application or supplement for BLI400 laxative, or, if the application is not approved, for two years after the drug investigation program is discontinued. These records will be made available at reasonable times for inspection and copying if requested by a properly authorized employee of Braintree Laboratories or the Department of Health and Human Services in accordance with federal regulations.

#### 13. PUBLICATION AND AGREEMENT

The results of this study will be published if mutually agreed by Braintree Laboratories and the Investigator and at a mutually agreed upon date. Investigator agrees to submit to Braintree Laboratories, within sixty (60) days of the proposed submission date, any proposed publication or presentation for prior review. Braintree Laboratories will, within thirty (30) days after receipt, advise if there is any proprietary or patentable information, which should not be disclosed at the present time. Investigator shall not release any such proposed publication or presentation, if so notified by Braintree Laboratories.

BLI400 (NDA 211281)

Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

#### 14. INVESTIGATORS AGREEMENT

I agree to perform the protocol according to Federal Regulations and as detailed in this document to the best of my ability. I recognize that if I fail to do so my participation in this study may be terminated. I also agree to the publication provisions stated in Section 13, above. My signature on the cover page of this protocol serves as documentation of my acceptance of the terms noted above.

BLI400 (NDA 211281)

Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

#### 15. REFERENCES

Drossman, D. (2000) Rome II: The Functional Gastrointestinal Disorders. Lawrence, KS: Allen Press.

Faruqui AA, Joshi, C. Lactitol: A Review of its Use in the Treatment of Constipation. International Journal of Recent Advances in Pharmaceutical Research 2012; 2(1): 1-5

Maydeo, A. Lactitol or lactulose in the treatment of chronic constipation: result of a systematic. <u>J Indian Med Assoc.</u> 2010;108(11):789-92.

Patil DH, Grimble GK, Silk DB. <u>Lactitol</u>, a new hydrogenated lactose derivative: <u>intestinal absorption and laxative threshold in normal human subjects</u>. Br J Nutr. 1987;57(2):195-9.

Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

## APPENDIX A

## Patient Assessment of Constipation – Quality of Life (PAC-QOL) Questionnaire

| 1 | |
|---|---|
| | PAC-QOL ® |
| | PATIENT ASSESSMENT OF CONSTIPATION |
| | The following questions are designed to measure the impact constipation has had on your daily life over the past 2 weeks. For each question, please check one box. |
| you<br>Du | The following questions ask about your symptoms related to constipation. During the past 2 weeks, to what extent or intensity have you Not at all of the past 2 weeks, to what extent or intensity have you A little bit of the past 2 weeks, to what extent or intensity have you A little bit of the past 2 weeks, to what extent or intensity have you |
| 1. | felt bloated to the point of bursting? |
| 2. | felt heavy because of your constipation? |
| Cor | The next few questions ask about how constipation affects your <u>daily life.</u> During the past 2 weeks, how much of the time the t |
| 3. | felt any physical discomfort? |
| 4. | felt the need to have a bowel movement but not been able to? |
| 5. | been embarrassed to be with other people? |
| 6. | been eating less and less because of<br>not being able to have bowel<br>movements? |

PAC-QOL

Copyright @ 1997. Janssen Research Foundation. All rights reserved.



Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

## Patient Assessment of Constipation – Quality of Life (PAC-QOL) Questionnaire

| The next few questions ask about how constipation affects your <u>daily life</u> . During the past 2 weeks, to what extent or intensity have you | | Not at all<br>0 | A little bit<br>1 | Moderately<br>2 | Quite a bit<br>3 | Extremely 4 |
|---|---|---|---|---|---|---|
| 7. | had to be careful about what you eat? | | | | | |
| 8. | had a decreased appetite? | | | | | |
| 9. | been worried about not being able to choose what you eat (for example, at a friend's house)? | | | | | |
| 10. | been embarrassed about staying in<br>the bathroom for so long when you<br>were away from home? | | | | | |
| 11. | been embarrassed about having to<br>go to the bathroom so often when<br>you were away from home? | | | | | |
| 12. | been worried about having to change<br>your daily routine (for example,<br>traveling, being away from home)? | | | | | |
| | • | | | | | |
| The next few questions ask about your feelings related to constipation. During the past 2 weeks, how much of the time have you | | None of<br>the time<br>0 | A little of<br>the time<br>1 | Some of<br>the time<br>2 | Most of<br>the time<br>3 | All of the<br>time<br>4 |
| 13. | felt irritable because of your condition? | | | | | |
| 14. | been upset by your condition? | | | | | |
| 15. | felt obsessed by your condition? | | | | | |
| 16. | felt stressed by your condition? | | | | | |
| 17. | felt less self-confident because of your condition? | | | | | |
| 18. | felt in control of your situation? | | | | | |

PAC-QOL

Copyright @ 1997. Janssen Research Foundation. All rights reserved.



Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

## Patient Assessment of Constipation – Quality of Life (PAC-QOL) Questionnaire

| The next questions ask about your<br>feelings related to constipation.<br>During the past 2 weeks, to what extent<br>or intensity have you | | Not at all<br>0 | A little bit<br>1 | Moderately<br>2 | Quite a bit<br>3 | Extremely<br>4 |
|---|---|---|---|---|---|---|
| 19. | been worried about not knowing<br>when you are going to be able to<br>have a bowel movement? | | | | | |
| 20. | been worried about not being able to have a bowel movement? | | | | | |
| 21. | been more and more bothered by not<br>being able to have a bowel<br>movement? | | | | | |
| with | next questions ask about your <u>life</u><br>neonstipation. During the past 2<br>eks, how much of the time have<br> | None of<br>the time<br>0 | A little of<br>the time<br>1 | Some of<br>the time<br>2 | Most of<br>the time<br>3 | All of the<br>time<br>4 |
| 22. | been worried that your condition will get worse? | | | | | |
| 23. | felt that your body was not working properly? | | | | | |
| 24. | had fewer bowel movements than you would like? | | | | | |
| deg | next questions ask about <u>your</u><br>ree of <u>satisfaction</u> related to<br>stipation. During the past 2 weeks, | | | | | |
| | hat extent or intensity have you | Not at all<br>0 | A little bit<br>1 | Moderately<br>2 | Quite a bit<br>3 | Extremely<br>4 |
| 25. | satisfied with how often you have a bowel movement? | | | | | |
| 26. | satisfied with the regularity of your bowel movements? | | | | | |
| 27. | satisfied with the time it takes for food to pass through the intestines? | | | | | |
| 28. | satisfied with your treatment? | | | | | |

PAC-QOL

Copyright @ 1997. Janssen Research Foundation. All rights reserved.



Braintree Laboratories, Inc. Protocol Number BLI400-303 Confidential

#### APPENDIX B

#### Patient Assessment of Constipation – Symptom (PAC-SYM) Questionnaire

#### Patient Assessment of Constipation-Symptom Questionnaire (PAC-SYM)

This questionnaire asks you about your constipation symptoms in the past two weeks. Answer each question according to your symptoms, as accurately as possible.

Please indicate how severe your symptoms have been during the past two weeks. If you have not had the symptom during the past two weeks, check 0. If the symptom seemed mild, check 1. If the symptom seemed moderate, check 2. If the symptom seemed severe, check 3. If the symptom seemed very severe, check 4. Please be sure to answer every question.

| How severe have each of these<br>symptoms been in the last two<br>weeks? | Absent<br>0 | Mild<br>1 | Moderate | Severe | Very<br>Severe<br>4 |
|---|---|---|---|---|---|
| discomfort in your abdomen | | | | | |
| 2. pain in your abdomen | | | | | |
| 3. bloating in your abdomen | | | | | |
| 4. stomach cramps | | | | | |
| 5. painful bowel movements | | | | | |
| rectal burning during or after a<br>bowel movement | | | | | |
| <ol><li>rectal bleeding or tearing during<br/>or after a bowel movement</li></ol> | ; | | | | |
| <ol> <li>incomplete bowel movement,<br/>like you didn't "finish"</li> </ol> | | | | | |
| <ol> <li>bowel movements that were too<br/>hard</li> </ol> | | | | | |
| bowel movements that were too<br>small | | | | | |
| straining or squeezing to try to<br>pass bowel movements | | | | | |
| feeling like you had to pass a bowel movement but you couldn't (false alarm) | | | | | |

Proprietary information of Janssen Research Foundation All rights reserved. 1997.
# An Open Label Study of Chronic Use of BLI400 Laxative in Constipated Adults

# **Braintree Protocol BLI400-303**

**Version Dated 4-13-2016** 

**SPONSOR** Braintree Laboratories, Inc.

60 Columbian St. West P.O. Box 850929 Braintree, MA 02185

PH: 781-843-2301

| Mark Cleveland | Date |
|------------------------------|------|
| Sr. Vice President, R&D/RA | |
| Braintree Laboratories, Inc. | |
| Principal Investigator | Date |

| 1. | INTRODUCTION | 5 |
|------------|--------------------------------------------------------|-------|
| 2. | STUDY OBJECTIVE | .10 |
| | STUDY PLAN | .10 |
| 3.1 | | |
| 3.2 | | |
| 3.3 | | |
| 3.4 | STUDY TREATMENTS | .10 |
| 3.5 | | .12 |
| | 3.5.1. Inclusion Criteria | |
| | 3.5.2. Exclusion Criteria | |
| 4. | STUDY PROCEDURES | |
| 4.1 | | .14 |
| | 4.1.1. Informed Consent | |
| | 4.1.2. Enrollment and Allocation of Subject Number | |
| | 4.1.3. Study Drug | 16 |
| | 4.2.1. Treatment Day 1 | . 1 ( |
| | 4.2.2. Visit 2 (Month 2) +/- 4 days | |
| | 4.2.3. Visit 3 (Month 4) +/- 4 days | |
| | 4.2.4. Visit 4 (Month 6) +/- 4 days | |
| | 4.2.5. Visit 5 (Month 9) +/- 4 days | |
| | 4.2.6. Visit 6 (Month 12 or Early Term) +/- 4 days | |
| 4.3 | 4.2.7. Follow-up Telephone Call (Day 374) +/- 4 days | 1.0 |
| 4.2 | | |
| 4.5 | | |
| 5. | ADVERSE EVENTS | .21 |
| 5.1 | . Adverse Event Definition and Reporting | .21 |
| 6. | SERIOUS ADVERSE EVENTS REPORTING | .23 |
| | INSTITUTIONAL REVIEW BOARD AND INFORMED CONSENT | _ |
| | MANAGEMENT OF INTERCURRENT EVENTS | |
| 8.1<br>8.2 | | |
| | DATA ANALYSIS | |
| 9.1<br>9.2 | | |
| 9.3 | | |
| | 9.3.1. Demographic and Baseline Characteristics25 | |
| | 9.3.2. Safety Analyses | |
| | 9.3.3. Efficacy Analyses (Patient Reported Outcomes)27 | |

| 9.4. | STUDY POPULATIONS | 27 |
|--------|-----------------------------------------------|----|
| 9.4.1. | Intention-to-Treat (ITT) Population | 27 |
| 9.4.1. | Modified Intention-to-Treat (mITT) Population | 27 |
| 9.4.2. | Per-Protocol Population | 28 |
| 10. DF | RUG INVENTORY AND DISPOSITION | 28 |
| 11. ST | UDY MONITORING | 28 |
| 12. DC | OCUMENTS AND NOTIFICATIONS | 28 |
| 12.1. | Informed Consent | 28 |
| 12.2. | Institutional Review Board | 28 |
| 12.3. | AMENDMENTS TO THE PROTOCOL | 29 |
| 12.4. | Data Records | 29 |
| 13. PU | UBLICATION AND AGREEMENT | 29 |
| 14. IN | VESTIGATORS AGREEMENT | 30 |
| 15. RE | EFERENCES | 31 |
| 16 AF | PPENDIX A | 32 |
| AF | PPENDIX B | |

#### CLINICAL PROTOCOL SUMMARY SHEET

#### STUDY TITLE:

An Open Label Study of Chronic Use of BLI400 Laxative in Constipated Adults

**PROTOCOL:** BLI400-303

**VERSION DATE:** 4-13-2016

**IND NUMBER:** 118,906

# **OBJECTIVE:**

To evaluate the safety of chronic use of BLI400 Laxative in constipated adults.

#### STUDY DESIGN:

This is an open-label, multi-center study in constipated outpatients.

#### **SUBJECTS:**

Approximately 300 male or female adult subjects with a history of constipation will be enrolled in this study (including approximately 100 elderly subjects).

#### **STUDY MEDICATIONS:**

BLI400 Laxative (21 grams of Lactitol Monohydrate, NF)

#### **DURATION OF TREATMENT**

Subjects will take BLI400 laxative daily for 12 months (52 weeks). Participation in this study will last for approximately 54 weeks, including the 14 day follow up telephone call.

## PRIMARY ENDPOINT

Safety will be analyzed through the use of adverse event and ECG data, and the comparison of chemistry, hematology, and urinalysis values as measured at baseline and at specific time points throughout the study.

#### 1. INTRODUCTION

The present approaches to the treatment of chronic idiopathic constipation (CIC) are limited and for some patients there are significant drawbacks that have not been resolved. It would be desirable to provide a source of relief for constipation that would permit dosing adjustments to optimize efficacy and safety and that would be pleasant to consume to improve patient compliance. The treatment should not have the safety issues associated with oral phosphate laxatives, have an acceptable safety profile, and be effective in numerous types of constipation.

Braintree Laboratories, Inc. is investigating the use of a new chemical composition, BLI400 (Lactitol Monohydrate NF Powder for Reconstitution) as a treatment for adult constipation. Ample published literature with lactitol provides significant preclinical and clinical studies which support the safe and effective use of this GRAS-listed compound.

These reports indicate that the BLI400 lactitol composition has promise as a candidate for further development for the treatment of constipation, as reviewed herein.

BLI400 is a member of the pharmaceutical class of osmotic laxatives; specifically it is a non-absorbed, colonically metabolized sugar alcohol (polyol). Studies reviewed here indicate it provides relief from the symptoms of constipation by rapidly inducing a patient-controlled bowel movement. While lactitol appears to be minimally, if at all, absorbed in the small intestine, colonic microbes split lactitol into D-galactose and D-sorbitol, which are fermentable to organic acids including lactic, formic, propionic, butyric and acetic acids (as reviewed in Patil et al, 1987). The osmotic properties of the small organic molecules consistently point to their pharmacodynamic effects as dependent on water retention with the stool. Thus, BLI400 is a pro-drug of an essentially non-absorbed osmotic laxative. Lactitol is generally considered to be pharmacologically inert and is often referred to as a "prebiotic" with no specific receptor targets for its laxative action.

#### Rationale for Performing Research with the Investigational Product

Lactitol monohydrate, at a daily dose of 21 grams per day appears to be a safe and effective treatment for constipation, but it has not been studied and proven in clinical

trials in the US. Lactitol appears to be a "prebiotic", a substrate for colonic bacteria which convert it into osmotically active small molecules. Extensive published and non-published literature supports its safety and efficacy, but a Phase III clinical trial is required for its registration in the US. It is envisaged there will be one, multi-site, controlled study in patients with documented constipation and that the design will be similar to other studies that have led to the approval of laxatives, such as those for MiraLAX, NDA 22-015 and consistent with FDA's recommendations for study endpoints in CIC trials.

#### Physical, Chemical, and Pharmaceutical Properties and Formulation

Lactitol is a simple monosaccharide sugar alcohol, a synthetic derivative of the milk sugar lactose that was discovered in the 1920s. It is a dry, free flowing powder, readily soluble in aqueous solutions. As shown by the structure diagrams, it is an analog of the disaccharide lactulose.

Lactitol

Lactulose

Table 1-1
Components of a Typical Single Dose of BLI400

| Component | Amount (g)* |
|--------------------------|-------------|
| Lactitol monohydrate, NF | 21 |

The product will be provided in multi-dose bottles with a measuring cap to deliver 10.5 grams of BLI400.

**Nonclinical Studies:** Extensive nonclinical studies have been performed with lactitol as support for its registration and marketing in countries outside the US and are reviewed in detail in the BLI400 Investigators' Brochure. The studies have covered basic pharmacology, genotoxicity and mutagenicity, acute and chronic studies including carcinogenicity and reproductive toxicity. These studies were carried out in mice, rats, dogs and rabbits.

**Pharmacology:** Lactitol is not degraded by the galactosidase enzymes of the small intestine However, colonic microflora degrade lactitol extensively in rats so that lactitol elevated the proportions of acetic acid and lowered proportions of butyric acid in the hindgut of rats. The osmotic effects of these organic acids appear to provide the pharmacodynamic basis for lactitol's laxative action. Increased output of moist feces was seen in all animals species studied in a dose-related manner. The highest doses tested caused frank diarrhea in some studies.

**Metabolic Effects:** In some studies, total serum cholesterol and triglycerides were reduced equally in rats fed diets containing 7% sorbitol or lactitol. By acidifying fecal contents, lactitol lowered ammonia levels in animal models of hepatic encephalopathy, perhaps as a result of production of the poorly absorbed ammonium ion that follows lowering the cecal pH. Rats fed a diet containing 5% of lactitol for two weeks displayed a significant increase of calcium absorption.

Toxicology Studies: Only weak edema ensued after lactitol application to intact skin, but erythema and edema emerged when it was applied to abraded skin. Rodents treated with lactitol had loose, frequent stools and cecal enlargement. This was often accompanied by decreased weight gain and increased water consumption. Clinical chemistry changes included changes in electrolyte levels, decreased cholesterol and alkaline phosphatase. Perhaps as compensation for the electrolyte changes that probably followed the diarrhea, adrenal weight and hypertrophy of the zona fasciculata were seen in the highest dose groups. Renal tubular degeneration with nephrocalcinosis was occasionally seen and may follow the increased calcium absorption. Lactitol was not considered positive for mutagenicity or chromosomal damage studied in standard in vitro and in vivo assays. Life-long carcinogenicity studies have indicated that Leydig cell dysplasia occurred in

rats at high lactitol doses, but this was not seen in mice dosed for 24 months or dogs dosed for 12 months. This species-specific effect in some rat strains was not considered significant to humans, since ordinary milk sugar, lactose, produces a similar effect in rodents.

Clinical Pharmacology and Safety: Since lactitol is extensively degraded to organic acids in the colon, it is little surprise that there are no published studies on its level in blood after administration. Some have estimated that only 0.6% of an oral dose of lactitol is excreted in urine. Similar to what is found in animals, lactitol is extensively metabolized in the human colon, making available a significant proportion of the metabolites for colonic absorption. Unlike in animals, lactitol does not seem to stimulate calcium absorption in humans, although in one study when 15 g of lactitol was administered along with calcium in solution to fasting volunteers, calcium absorption was diminished. Administering lactitol increases fecal Bifidobacteria levels, while other bacteria (fecal anaerobes, aerobes, Enterobacteriaceae or lactobacilli) were unaffected. After the ingestion of 25 g lactitol, xylitol, or glucose by eight healthy male volunteers the rise in plasma glucose was significantly greater 30 and 60 minutes after ingestion of glucose while no rise in plasma glucose followed ingestion of lactitol.

The investigation of the use of a mixture of lactitol for the treatment of constipation has been extensively studied, but the information is only available in published form. From these observations, it appears that lactitol's adverse events are limited largely to the gastrointestinal system. Symptoms such as nausea, cramps, abdominal pain, flatulence and vomiting may be expected and could lead to withdrawal from the study if not controlled. Their incidence and severity may be ameliorated in some patients by dose-adjustment. Changes in hematology, clinical chemistry or urinalysis may be seen, and their clinical significance will be assessed during the development of lactitol. In one study plasma potassium was elevated with lactitol, but the values stayed within the normal range.

Clinical Efficacy: Lactitol has been marketed since at least 1985 outside the US in Europe and other regions (where it is known as Lactitol Ex-Lax® or Importal®, for example) as a syrup or powder for the treatment of constipation in adults, including the elderly and children. As a result a substantial body of evidence has accumulated on its

use in treating constipation, as evidenced by more than 19 publications since 1988, including two recent review articles (Maydeo, 2010; Faruqui and Joshi, 2012).

A minimal effective dose of 0.25 g/kg has been suggested, and most studies have found that a starting dose of 20 g of lactitol is effective and produces minimal side effects. Some studies that have allowed the subjects to make dosage increases to achieve relief of constipation symptoms and dose reductions to minimize side effects have indicated that this strategy can optimize therapy.

Maydeo (2010) presented a systematic review of six published randomized, non-randomized and open trials comparing the safety and efficacy of lactitol to those of lactulose. Overall, lactitol was comparable to lactulose in efficacy measures (normal stool consistency and number of bowel movement per week). Patients found lactitol to be more acceptable and were more compliant with it largely due to its superior palatability (73.2 % vs. 26.8 %). Lactitol was significantly better than lactulose in the frequency of adverse events (31.2  $\pm$  0.8 % vs. 62.1  $\pm$ 1.1 %, p= 0.0019). The physicians' assessment favored lactitol as compared to lactulose (61.91% vs. 47.83%). The following table is adapted from Maydeo's summary of the reviewed trials.

| Parameter Evaluated | Lactitol | Lactulose |
|--------------------------------------|------------------|------------------|
| Patient's acceptance | 73.2% | 26.8% |
| Consistency of stool (normal/soft) | $80.5 \pm 4.5\%$ | $75.0 \pm 8.0\%$ |
| Bowel movement/week | $5.9 \pm 0.2$ | $5.6 \pm 0.6$ |
| Incidence of side-effects | $31.2 \pm 0.8$ | 62.1 ±1.1% |
| Global efficacy judged by physicians | 61.9% | 47.8% |

#### 2. STUDY OBJECTIVE

To evaluate the safety of chronic use of BLI400 laxative in constipated adults.

#### 3. STUDY PLAN

#### 3.1. Study Design

This is an open-label, multi-center study in which constipated subjects will receive BLI400 for 12 months.

# 3.2. Number of Subjects

Approximately 300 constipated subjects will be enrolled into this study, including approximately 100 elderly subjects ( $\geq$  65 years of age at Visit 1).

#### 3.3. **Duration of Study**

Qualifying subjects will receive BLI400 at Visit 1 and will begin a 12-month Treatment Period. Subjects will return for clinic visits at the end of Months 2, 4, 6, 9 and 12. A follow up call will take place 2 weeks after the end of treatment. A completed subject is defined as a subject that completes the Visit 6 (Month 12) visit.

#### 3.4. Study Treatments

## **BLI400 Laxative**

BLI400 laxative will be provided polyethylene bottles containing sufficient study medication for 30 days of dosing. The bottles will be equipped with a cap that can be used to measure 10.5 grams of BLI400. Each bottle will also have a clinical label containing a caution statement, study code, study sponsor and subject number. Subjects will be instructed to mix the contents of 2 capfuls (approximately 21 g) in 4 - 8 oz of juice or other beverage, and take once daily preferably in the morning. Subjects that develop persistent diarrhea or loose stools will be allowed to adjust their dose down to 10.5g (1 capful) per day.

## **Rescue Bisacodyl**

Subjects will be dispensed bisacodyl at each study visit (previously dispensed bisacodyl may be redispensed if needed, although this is not encouraged). Subjects will be instructed to take 5 - 10 mg (1 - 2 tablets) of bisacodyl if they are experiencing severe discomfort due to their constipation, or have not had a BM in 4 days. No more than 6 tablets (30mg) of bisacodyl should be taken in a week.

If a subject does not have a bowel movement within 24 hours of taking a bisacodyl dose, a second dose should be taken. If after the second bisacodyl dose the subject does not have a BM within 24 hours, the subject should contact the site. The investigator should then consider having the subject return for an evaluation and/or discontinuing the subject from the study.

All study medication is required to remain at room temperature 20°-25°C (68°-77°F); excursions permitted between 15°-30°C (59°-86°F).

# 3.5. Subject Selection

#### 3.5.1. Inclusion Criteria

Subjects will be admitted to the study if they are:

- 1. Male or female subjects at least 18 years of age
- 2. Constipated, defined by the following adapted ROME II definition (Drossman et al, 2000):
  - A. Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for at least 12 weeks (which need not be consecutive) in the preceding 12 months:
    - a. Straining during > 25% of defecations
    - b. Lumpy or hard stools in > 25% of defecations
    - c. Sensation of incomplete evacuation for > 25% of defecations
- 3. If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, sterilized, abstinent, or vasectomized spouse)
- 4. Negative urine pregnancy test at screening, if applicable
- 5. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

#### 3.5.2. Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

- 1. Report loose (mushy) or water stools in the absence of laxative use for more than 25% of BMs during the 12 weeks before Visit 1
- 2. Meet the Rome II criteria for Irritable Bowel Syndrome: reports abdominal discomfort or pain that has two or more of the following three features for at least 12 weeks, which need not be consecutive, in the 12 months before Visit 1:
  - Relieved with defecation
  - Onset associated with a change in frequency of stool
  - Onset associated with a change in form (appearance of stool)
- 3. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
- 4. Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
- 5. Subjects with hypothyroidism that is being treated and for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of Visit 1
- 6. Subjects taking laxatives, enemas or prokinetic agents that refuse to discontinue these treatments from Visit 1 until after completion of Visit 6
- 7. Subjects who are pregnant or lactating, or intend to become pregnant during the study
- 8. Subjects of childbearing potential who refuse a pregnancy test
- 9. Subjects who are allergic to any BLI400 component (lactitol)
- 10. Subjects taking narcotic analysesics or other medications known to cause constipation.
- 11. Subjects with clinically significant cardiac abnormalities identified at the Visit 1 ECG
- 12. Subjects with clinically significant laboratory abnormalities, deemed as a potential safety issue by the Investigator, may be discontinued at the Investigator's discretion.
- 13. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
- 14. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
- 15. Subjects with an active history of drug or alcohol abuse
- 16. Subjects have been hospitalized for a psychiatric condition or have made a suicide attempt during the 2 years before Visit 1
- 17. Subjects who withdraw consent at any time prior to completion of Visit 1 procedures

#### 4. STUDY PROCEDURES

Study procedures are described as follows and depicted graphically in Section 4.3, below. Acceptable deviations from the visit schedule are indicated. These variations must not be cumulative; i.e. visits should always be scheduled in relationship to Visit 1 (Day 0).

## 4.1. Visit 1 (Day 0)

At the screening visit, the following procedures will be undertaken:

- Subject is fully informed about the study and gives written agreement to study participation in the form of a signed informed consent form (refer to Section 4.1.1)
- Assess eligibility (refer to inclusion/exclusion criteria)
- Review of medications
- Medical history including history of constipation (ROME criteria See Inclusion #2)
- Physical examination
- Vital signs, including assessment of orthostatic hypotension (while seated and after standing for a minimum of 2 minutes) including height and bodyweight, pulse and temperature
- A 12-lead ECG will be performed by qualified, trained site personnel. ECG output must be reviewed by a physician investigator. Any clinically significant cardiac abnormalities identified on the ECG should disqualify a subject. Data from the ECG will be collected in the eCRF.
- Urine pregnancy test (if applicable)
- Blood and urine samples will be collected for testing at a central laboratory, as shown below.

<u>Chemistry:</u> alkaline phosphatase, ALT, anion gap, AST, bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatine kinase, creatinine, eGFR, GGT, HCG, inorganic phosphate, magnesium, osmolality, potassium, sodium, uric acid. CK-MB will be tested in samples where the CK value is greater than 2.5 times the upper normal limit.

<u>Hematology:</u> hematocrit, hemoglobin, platelets count, red blood cell count, white blood cell count (and differentials)

<u>Urinalysis:</u> including electrolytes (sodium, potassium, magnesium, calcium), microscopic analysis, urine osmolality

Subjects with clinically significant laboratory abnormalities, deemed as a potential safety issue by the Investigator, may be discontinued at the Investigator's discretion.

If the subject is eligible for the study, assign a subject number.

 Subjects will complete the Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL, refer to Appendix A) and the Patient Assessment of Constipation Symptom questionnaire (PAC-SYM, refer to Appendix B)

- Dispense 2 bottles of BLI400
- Dispense rescue bisacodyl. Subjects will be allowed to take 5 10mg of bisacodyl if they
  are experiencing severe discomfort due to their constipation, or have not had a BM in 4
  days.
- Instruct subject to maintain their normal dietary habits during study participation
- Schedule the next study visit to occur after 60 days

Subjects that are ineligible due to prohibited medication use (Exclusion Criterion 10) may be washed out for a period of 14 days. No additional procedures should be performed on these subjects. After the washout period, subjects may be enrolled and all Visit 1 procedures should be repeated (with the exception of obtaining informed consent).

#### 4.1.1. Informed Consent

Following the informed consent process, study subjects will sign a current IRB approved consent form. No study procedures may be performed prior to the subject providing informed consent. The subject's original signed and personally dated Informed Consent Form (together with any subsequent IRB approved amended versions) must be retained by the Investigator in the subject's file. A copy of the original signed and dated Informed Consent Form must be given to the subject.

#### 4.1.2. Enrollment and Allocation of Subject Number

Subjects will be enrolled into the study only when they have given their written, informed consent to participate.

Subjects enrolled at the screening visit will be assigned a subject number by site personnel.

This number will consist of:

- The 3-digit Site Number;
- The 3-digit subject identifier number (this number is a sequentially allocated number). Each site will begin with 001 for the first subject screened, 002 for the second and so on. For example, the third subject screened at Site 15 will become Subject Number 15-003. After a subject completes all screening procedures and eligibility has been confirmed, site personnel will assign a subject number.

#### 4.1.3. Study Drug

After it has been confirmed that all eligibility criteria have been met, site personnel will utilize the IWRS to assign a drug kit number to the subject.

Site personnel must only dispense the drug kit that has been assigned by the IWRS. Dispensing of incorrect kits is considered a protocol violation.

Subjects will be provided instructions on how to take the study medication and rescue medication. Two bottles will be dispensed per subject. The study drug bottles will be weighed for drug accountability purposes. Subjects will be instructed to return all bottles at each follow up visit.

#### 4.2. Treatment Period

#### 4.2.1. Treatment Day 1

Starting on the morning of Treatment Day 1 (the day after Visit 1), subjects will measure 2 capfuls of study medication and ingest it mixed in a beverage of their choice. Subject will take a daily dose of 2 capfuls until they return for Visit 2. Subjects that develop persistent diarrhea or loose stools should contact their study center. These subjects will be allowed to adjust their dose down to 10.5g (1 capful) per day.

#### 4.2.2. Visit 2 (Month 2) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 2 (Day 60). Vital signs (see section 4.1 for details) and ECGs will be recorded. Study personnel will weigh returned bottles and count rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Subjects will be dispensed 2 new bottles of study medication. Subjects will be instructed to return all bottles and bisacodyl at the next follow up visit.

#### 4.2.3. Visit 3 (Month 4) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 3 (Day 120). Vital signs (See section 4.1 for details) will be recorded. Study personnel will weigh returned bottles and count rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications.

Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Subjects will be dispensed 2 new bottles of study medication. Subjects will be instructed to return all bottles and bisacodyl at the next follow up visit.

## 4.2.4. Visit 4 (Month 6) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 4 (Day 180). Vital signs (See section 4.1 for details) will be recorded. Study personnel will review returned bottles and rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Subjects will be dispensed 3 new bottles of study medication. Subjects will be instructed to return all bottles and bisacodyl at the next follow up visit.

## 4.2.5. Visit 5 (Month 9) +/- 4 days

Subjects will continue to take BLI400 daily and will return to the clinic for Visit 5 (Day 270). Vital signs (See section 4.1 for details) will be recorded. Study personnel will review returned bottles and rescue bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section 4.1. Three new bottles of study medication will be dispensed at this visit. Subjects will be instructed to return all bottles and bisacodyl at Visit 6.

#### 4.2.6. Visit 6 (Month 12 or Early Term) +/- 4 days

Subjects will return at Day 360 for their final clinic visit. Vital signs (see section 4.1 for details) and ECGs will be recorded. A physical examination will be performed. Study personnel will weigh returned bottles and count bisacodyl for accountability purposes. Subjects will be queried for any adverse events or changes to their concomitant medications. Subjects will complete the PAC-QOL and PAC-SYM questionnaires. Samples for chemistry, hematology and urinalysis will be repeated as outlined in Section

4.1. Clinically significant laboratory abnormalities present at Visit 6 should be followed until resolved or are considered stable.

# 4.2.7. Follow-up Telephone Call (Day 374) +/- 4 days

At Day 374, approximately 2 weeks after the last study visit or early term visit, site personnel will contact subjects by telephone to query if any new adverse events have occurred and if any adverse events ongoing at Visit 6 have resolved. Subjects will also be asked about the status of their concomitant medications.

# 4.3. Tabulated Study Procedures

The following graphically depicts the flow of study procedures at each visit.

| Procedures | Visit 1<br>Day 0 | Visit 2<br>Month 2 | Visit 3<br>Month 4 | Visit 4<br>Month 6 | Visit 5<br>Month 9 | Visit 6<br>Month 12/<br>ET | <b>☎</b> Day 374 +/- 4 days |
|---|---|---|---|---|---|---|---|
| | | +/- 4 days | +/- 4 days | +/- 4 days | +/- 4 days | +/- 4 days | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria Review | X | | | | | | |
| Medical History | X | | | | | | |
| Physical Examination | X | | | | | X | |
| Vital Signs <sup>1</sup> | X | X | X | X | X | X | |
| Electrocardiogram | X | X | | | | X | |
| Review of Concomitant Medication | X | X | X | X | X | X | X |
| Urine Pregnancy Test (if applicable) <sup>2</sup> | X | | | | | | |
| Enroll Eligible Subjects | X | | | | | | |
| Subject to Complete PAC-QOL, PAC-SYM | X | X | X | X | X | X | |
| Blood Sample for Chemistry Testing | X | X | X | X | X | X | |
| Blood Sample for Hematology Testing | X | X | X | X | X | X | |
| Urine Sample for Urinalysis | X | X | X | X | X | X | |
| Blood Sample for Serum Pregnancy Testing | | | | X | | X | |
| Dispense Study Drug and Rescue Bisacodyl | X | X | X | X | X | _ | |
| Study Drug and Rescue Bisacodyl Accountability | | X | X | X | X | X | |
| Assess Safety | | X | X | X | X | X | X |

blood pressure and pulse while seated and after standing for 2 minutes, temperature, weight and height (@Visit 1 only)

<sup>&</sup>lt;sup>2</sup>refer to Section 4.4

## 4.4. Pregnancy

Subjects who are female and of childbearing potential must have a urine pregnancy test done at screening. A positive result will rule out the participation of the subject in the study. Serum pregnancy tests will be performed at Visits 4 (Month 6) and 6 (Month 12). If a subject becomes pregnant during the study, the subject must be removed from the study and followed until one month after the end of the pregnancy.

Female study subjects must be surgically sterilized or using oral contraceptives, depot contraceptives, double-barrier method, intrauterine device, or testifies that she is monogamous with a vasectomized partner. Subjects practicing abstinence must agree to use an acceptable form of birth control should they become sexually active during the study.

Women with a history of bilateral tubal ligation are not considered of childbearing potential and are not required to have a urine pregnancy test at screening.

Oral contraceptives, hormone implants, and injections are only considered effective if started at least 1 month before the study.

Menopausal status is defined when menses have been absent for 12 months in a woman of appropriate age (usually 45 to 55 years) who has no other suspected or identified cause of amenorrhea.

#### 4.5. Concomitant Medications

The use of concomitant medication will be recorded from 7 days prior to Visit 1 until the end of the study at the telephone contact on Day 374. Subjects enrolled in this study will not be permitted to take any laxatives (other than the sponsor supplied rescue bisacodyl), whether prescription or over-the-counter, from Visit 1 until after completion of Visit 6. Any restricted laxative use during the study may result in termination of subject's participation. Subjects may not initiate treatment with any constipating medication.

#### 5. **ADVERSE EVENTS**

#### 5.1. Adverse Event Definition and Reporting

An Adverse Event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product.

Adverse event collection will coincide with the subject providing informed consent to participate in the study and will conclude with the end of study participation at Day 374 Follow-up Call. Diarrhea should be reported as an adverse event if a subject has more than 3 watery stools per day. Subjects with clinically significant laboratory results at Visit 6 which are classified by the Investigator as adverse events should return for a repeat blood draw. Subjects will be instructed to report promptly adverse events to the Investigator. The Investigator will record date/time of report, date/time of onset, description of the adverse event, severity of adverse event, action(s) taken regarding treatment of the event, action(s) taken regarding study participation, duration of adverse event, and the Investigator's assessment of relationship of adverse event to study treatment.

The Investigator should assess the severity of each adverse event using the following categories:

| Grade | Severity | Description |
|---|---|---|
| 1 | Mild | Barely noticeable, does not influence functioning |
| | IVIIIU | Causing no limitations of usual activities |
| 2 | Moderate | Makes participant uncomfortable, influences functioning |
| Moderate | | Causing some limitations of usual activities |
| 3 | | Severe discomfort, treatment needed |
| | Severe | Severe and undesirable, causing inability to carry out usual |
| | | activities |
| 4 | Life | Immediate risk of death |
| | threatening | Life threatening or disabling |
| 5 | Fatal | Causes death of the participant |

The Investigator should assess the relationship to study drug for each adverse event using the following categories:

| Categories of Attribution: | Description |
|---|---|
| UNRELATED | There is <i>no</i> evidence of any causal relationship. |
| POSSIBLE | There is <i>some</i> evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, the influence of <i>other factors may have contributed</i> to the event (e.g., the patient's clinical condition, other concomitant events). |
| PROBABLE | There <i>is evidence</i> to suggest a causal relationship, and the influence of other factors is <i>unlikely</i> . |
| DEFINITE | There is <i>clear</i> evidence to suggest a causal relationship, and other possible contributing factors can be <i>ruled out</i> . |

In published Phase 3 studies, adverse events associated with BLI400 administered at doses required for effective treatment of constipation included flatulence, nausea, vomiting, abdominal cramping or pain and bloating. These adverse reactions were transient and subsided rapidly upon dose adjustment or cessation.

#### 6. SERIOUS ADVERSE EVENTS REPORTING

A Serious Adverse Event (SAE) is any untoward medical occurrence that results in at least one of the following outcomes:

- Results in death
- Is life-threatening
- Requires inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly/birth defect
- Requires medical or surgical intervention to prevent permanent impairment or damage

SAE collection will coincide with the subject providing informed consent to participate in the study and will conclude 30 days after a subject's last dose of study medication. Should a serious and/or unexpected adverse event occur, the Investigator must notify Braintree Laboratories immediately. The Investigator will make a decision regarding continuing the subject's study participation, and may request input from Braintree Laboratories. The Investigator will be responsible for recommending or providing the subject with appropriate medical therapy. All subjects experiencing serious adverse events will be followed until satisfactory resolution occurs. Braintree Laboratories must be kept apprised of all follow-ups relative to serious adverse events. In addition, Investigators must comply with the SAE reporting requirements of the Institutional Review Board with oversight of the study.

Any serious and/or unexpected adverse events that occur during the study will be reported to Braintree Laboratories as follows:

Contact Telephone Numbers:

During Business hours

(M-F, 8:30 am - 5:00 pm EDT)

After hours or weekends



Braintree Laboratories and its medical monitor will review the report and determine whether an FDA Form 3500A will also be completed and sent to FDA.

#### 7. INSTITUTIONAL REVIEW BOARD AND INFORMED CONSENT

Institutional Review Board (IRB) review and approval of the study protocol and Informed Consent Form will be obtained prior to initiation of the study. Amendments to the study protocol and consent form generated during the course of the study will also require IRB approval.

#### 8. MANAGEMENT OF INTERCURRENT EVENTS

#### 8.1. Modification of Protocol

Neither an Investigator nor Braintree Laboratories will modify the protocol without first obtaining the concurrence of the other and the IRB. Investigators that continually violate the protocol or commit a serious violation may be subject to termination from the study. The study may be halted if at any time an Investigator or Braintree Laboratories deems the incidence or severity of adverse events to be unacceptable.

#### 8.2. Subjects Discontinued from the Study

Subjects may be dropped from the study for any of the following reasons:

- 1) Subject took prohibited medications during the Treatment Period
- 2) An adverse event requiring discontinuation (including failure to tolerate study medication).
- 3) The Investigator decides that the subject should be dropped from the study (e.g. serious adverse event, protocol violation, non-compliance).
- 4) The subject decides to withdraw from the study. Subjects are free to withdraw their consent and discontinue participation in the study at any time.

Braintree Laboratories should be contacted if possible prior to discontinuation of any subject. If a subject is discontinued from the study, Braintree Laboratories must be notified with an explanation for all discontinuances.

#### 9. DATA ANALYSIS

# 9.1. Sample Size

Consistent with ICH E1A Guideline for Industry, the Extent of Population Exposure to Assess Clinical Safety: for Drugs Intended for Long-term Treatment of Non-Life-Threatening Conditions (March 1995), 300 subjects will be treated with BLI400 for 12 months. This will allow for detection of adverse events that may increase in frequency or severity over time.

#### 9.2. Parameters to be Analyzed

The primary objective of this study is to investigate the safety of BLI400 used chronically for 12 months in subjects with constipation. Safety will be analyzed using ECG, vital signs, chemistry, hematology and urinalysis and adverse event data. Treatment emergent adverse event rates will be descriptively presented by preferred term, severity, and relationship to treatment.

# 9.3. Planned Analyses

#### 9.3.1. Demographic and Baseline Characteristics

Baseline demographic characteristics will be tabulated with N, mean, standard deviation, and range of values where appropriate

- Age
- Gender
- Race/ethnicity
- Constipation History

#### 9.3.2. Safety Analyses

Analysis of safety will be performed using the modified Intent to Treat population (see Section 9.4).

#### Adverse Events

Adverse Events will be coded using the MedDRA classification to provide a preferred term and primary system organ class for each event. Proportions of subjects with adverse events will be presented for the overall study population, and each demographic subgroup (age, gender and race). Tables of AEs will be presented by system organ class and preferred term, and include overall totals for AEs within each system organ class. Counting will be done by subject and not by event. A table of counts and percentages will also be made of those subjects with SAEs or AEs which led to withdrawal from the study.

Treatment-emergent AEs are defined as adverse events that had an onset day and time on or after the day and time of the first dose of study drug until the Day 374 Follow-up Call. Adverse Events having missing onset dates will be considered as treatment emergent.

The difference in adverse event rates between study periods will be tested by Chi-Square or Fisher's exact test with 95% confidence intervals.

## Laboratory Parameters

Summary statistics (i.e., mean, minimum, maximum, standard deviation, and number of subjects) will be presented for each laboratory parameter at each visit. Laboratory data will be summarized for the overall population and the elderly and non-elderly subgroups. When calculating the summary statistics only, the last observation within a visit window will be used if there are multiple observations. Changes from baseline (Visit 1) will be presented in a similar format. An additional listing will be provided of those subjects who have clinically significant laboratory values. The data will also be presented as shift tables and clinically significant abnormalities will be examined.

Results of laboratory tests for the change from baseline (Visit 1) and group differences will be tested using ANOVA.

#### Vital Signs

Summary statistics (i.e., mean, minimum, maximum, standard deviation, and number of subjects) will be presented for each vital sign at each visit and compared to the values obtained at Visit 1. When calculating the summary statistics only, the last observation within a visit window will be used if there are multiple observations. The data will also be presented as shift tables and clinically significant abnormalities will be examined.

ECG variables will be tabulated and presented for data collected at each visit. Data will be tabulated and summarized with descriptive statistics (N, mean, SD, CV%, SEM, minimum, and maximum) for each of the ECG variables. The differences in ECG variables between Visit 1 (Baseline), Visit 2 and Visit 6 will be tested using ANOVA.

## 9.3.3. Efficacy Analyses (Patient Reported Outcomes)

Subject constipation symptoms and quality of life indicators will be analyzed using data from the subject-completed PAC-SYM and PAC-QOL instruments. Change from baseline to each visit time point will be presented for each collected measure and will be tested using ANOVA. Data for each measure and time point will also be presented categorically by severity and tested using Chi-Square or Fisher's exact test.

#### 9.4. Study Populations

The following populations have been defined for data analyses.

#### 9.4.1.Intention-to-Treat (ITT) Population

This population includes all enrolled subjects that were dispensed study medication.

#### 9.4.1. Modified Intention-to-Treat (mITT) Population

This population consists of all enrolled subjects that took at least one dose of study medication. This population will be utilized for all safety analyses.

# 9.4.2. **Per-Protocol Population**

The per-protocol (PP) population will consist of all subjects in the mITT population who have not violated study entry criteria and have not deviated significantly from the protocol during the course of the study. Any analyses from this population will be considered as supportive to the ITT and mITT analyses. Reasons for exclusion from the PP population will be defined in the clinical study report.

#### 10. DRUG INVENTORY AND DISPOSITION

At the conclusion of the study, all drug materials will be accounted for. Federal law requires that, at the conclusion of the study, all drug materials must be returned to the study sponsor or destroyed according to local regulations.

#### 11. STUDY MONITORING

A Braintree Laboratories Study Monitor or qualified designee will visit the study center prior to the commencement of the study and periodically during the course of the study in accordance with federal guidelines governing the sponsorship of studies.

#### 12. DOCUMENTS AND NOTIFICATIONS

#### 12.1. Informed Consent

Written informed consent will be obtained from the subjects by the Investigator and will be kept on file at the study center. Documentation of the consent process should be noted in the study source documents.

#### 12.2. Institutional Review Board

Peer review and approval of the protocol by an appropriate Institutional Review Board is required prior to commencement of enrollment. Amendments to the approved protocol must also be submitted to the Institutional Review Board and approved prior to their implementation.

#### 12.3. Amendments to the Protocol

The Investigator and Braintree Laboratories will discuss any amendments to the study protocol. If an agreement is reached regarding the need for the amendment, it will be produced in writing by Braintree Laboratories and will be made a formal part of the protocol only after approval by an Institutional Review Board.

#### 12.4. Data Records

Site personnel will be required to enter study data into electronic case report forms (eCRFs) provided by Braintree Laboratories. Subject medical records will be reviewed to verify study data points, including potential adverse events, and to ensure correctness and consistency with the CRF entries. The Investigator should retain copies of paper and electronic data, patient consent/assent forms, and other study documents for a period of two years following the date of approval of a New Drug Application or supplement for BLI400 laxative, or, if the application is not approved, for two years after the drug investigation program is discontinued. These records will be made available at reasonable times for inspection and copying if requested by a properly authorized employee of Braintree Laboratories or the Department of Health and Human Services in accordance with federal regulations.

#### 13. PUBLICATION AND AGREEMENT

The results of this study will be published if mutually agreed by Braintree Laboratories and the Investigator and at a mutually agreed upon date. Investigator agrees to submit to Braintree Laboratories, within sixty (60) days of the proposed submission date, any proposed publication or presentation for prior review. Braintree Laboratories will, within thirty (30) days after receipt, advise if there is any proprietary or patentable information, which should not be disclosed at the present time. Investigator shall not release any such proposed publication or presentation, if so notified by Braintree Laboratories.

# 14. INVESTIGATORS AGREEMENT

I agree to perform the protocol according to Federal Regulations and as detailed in this document to the best of my ability. I recognize that if I fail to do so my participation in this study may be terminated. I also agree to the publication provisions stated in Section 13, above. My signature on the cover page of this protocol serves as documentation of my acceptance of the terms noted above.

#### 15. REFERENCES

Drossman, D. (2000) Rome II: The Functional Gastrointestinal Disorders. Lawrence, KS: Allen Press.

Faruqui AA, Joshi, C. Lactitol: A Review of its Use in the Treatment of Constipation. International Journal of Recent Advances in Pharmaceutical Research 2012; 2(1): 1-5

Maydeo, A. Lactitol or lactulose in the treatment of chronic constipation: result of a systematic. <u>J Indian Med Assoc.</u> 2010;108(11):789-92.

Patil DH, Grimble GK, Silk DB. <u>Lactitol</u>, a new hydrogenated lactose derivative: <u>intestinal absorption and laxative threshold in normal human subjects.</u> Br J Nutr. 1987;57(2):195-9.

# APPENDIX A

# Patient Assessment of Constipation – Quality of Life (PAC-QOL) Questionnaire

| | PAC-QOL ® |
|---|---|
| | PATIENT ASSESSMENT OF CONSTIPATION |
| | The following questions are designed to measure the impact constipation has had on your daily life over the past 2 weeks. For each question, please check one box. |
| you<br>Dur | The following questions ask about your symptoms related to constipation. During the past 2 weeks, to what extent or intensity have you Not at all 0 1 2 3 4 |
| 1. | felt bloated to the point of bursting? |
| 2. | felt heavy because of your constipation? |
| con<br>Dur | The next few questions ask about how constipation affects your <u>daily life</u> . None of A little of Some of Most of All of the time |
| 3. | felt any physical discomfort? |
| 4. | felt the need to have a bowel movement but not been able to? |
| 5. | been embarrassed to be with other people? |
| 6. | been eating less and less because of<br>not being able to have bowel<br>movements? |

Copyright @ 1997. Janssen Research Foundation. All rights reserved.



Г

# Patient Assessment of Constipation – Quality of Life (PAC-QOL) Questionnaire

| Cor | e next few questions ask about how<br>nstipation affects your <u>daily life</u> .<br>ring the past 2 weeks, to what extent<br>ntensity have you | Not at all<br>0 | A little bit<br>1 | Moderately<br>2 | Quite a bit<br>3 | Extremely<br>4 |
|---|---|---|---|---|---|---|
| 7. | had to be careful about what you eat? | | | | | |
| 8. | had a decreased appetite? | | | | | |
| 9. | been worried about not being able to<br>choose what you eat (for example, at<br>a friend's house)? | | | | | |
| 10. | been embarrassed about staying in<br>the bathroom for so long when you<br>were away from home? | | | | | |
| 11. | been embarrassed about having to<br>go to the bathroom so often when<br>you were away from home? | | | | | |
| 12. | been worried about having to change<br>your daily routine (for example,<br>traveling, being away from home)? | | | | | |
| <u> </u> | | | | | | |
| fee<br>Du | e next few questions ask about your<br>lings related to constipation.<br>ring the past 2 weeks, how much of<br>time have you | None of<br>the time<br>0 | A little of<br>the time<br>1 | Some of<br>the time<br>2 | Most of<br>the time<br>3 | All of the<br>time<br>4 |
| 13. | felt irritable because of your condition? | | | | | |
| 14. | been upset by your condition? | | | | | |
| 15. | felt obsessed by your condition? | | | | | |
| 16. | felt stressed by your condition? | | | | | |
| 17. | felt less self-confident because of your condition? | | | | | |
| 18. | felt in control of your situation? | | | | | |

PAC-QOL

Copyright @ 1997. Janssen Research Foundation. All rights reserved.

+

| <u>feel</u><br>Dur | next questions ask about your<br>ings related to constipation.<br>ing the past 2 weeks, to what extent<br>ntensity have you | Not at all<br>0 | A little bit | Moderately<br>2 | Quite a bit | Extremely<br>4 |
|---|---|---|---|---|---|---|
| 19. | been worried about not knowing<br>when you are going to be able to<br>have a bowel movement? | | | | | |
| 20. | been worried about not being able to have a bowel movement? | | | | | |
| 21. | been more and more bothered by not<br>being able to have a bowel<br>movement? | | | | | |
| with | next questions ask about your <u>life</u><br>neonstipation. During the past 2<br>eks, how much of the time have<br> | None of<br>the time<br>0 | A little of<br>the time<br>1 | Some of<br>the time<br>2 | Most of<br>the time<br>3 | All of the<br>time<br>4 |
| 22. | been worried that your condition will get worse? | | | | | |
| 23. | felt that your body was not working properly? | | | | | |
| 24. | had fewer bowel movements than you would like? | | | | | |
| Ь— | | | | | | |
| deg | next questions ask about <u>your</u><br>ree of satisfaction related to<br>stipation. During the past 2 weeks, | | | | | |
| | hat extent or intensity have you | Not at all<br>0 | A little bit<br>1 | Moderately<br>2 | Quite a bit<br>3 | Extremely<br>4 |
| 25. | satisfied with how often you have a bowel movement? | | | | | |
| 26. | satisfied with the regularity of your bowel movements? | | | | | |
| 27. | satisfied with the time it takes for food to pass through the intestines? | | | | | |
| 28. | satisfied with your treatment? | | | | | |

| PAC-QOL | |
|---------|---------|
| | PAC-QOL |

Copyright @ 1997. Janssen Research Foundation. All rights reserved.



APPENDIX B

# Patient Assessment of Constipation – Symptom (PAC-SYM) Questionnaire

## Patient Assessment of Constipation-Symptom Questionnaire (PAC-SYM)

This questionnaire asks you about your constipation symptoms in the past two weeks. Answer each question according to your symptoms, as accurately as possible.

Please indicate how severe your symptoms have been during the past two weeks. If you have not had the symptom during the past two weeks, check 0. If the symptom seemed mild, check 1. If the symptom seemed moderate, check 2. If the symptom seemed severe, check 3. If the symptom seemed very severe, check 4. Please be sure to answer every question.

| How severe have each of these<br>symptoms been in the last two<br>weeks? | | Absent<br>0 | Mild<br>1 | Moderate<br>2 | Severe<br>3 | Very<br>Severe<br>4 |
|---|---|---|---|---|---|---|
| 1. | discomfort in your abdomen | | | | | |
| 2. | pain in your abdomen | | | | | |
| 3. | bloating in your abdomen | | | | | |
| 4. | stomach cramps | | | | | |
| 5. | painful bowel movements | | | | | |
| | rectal burning during or after a<br>bowel movement | | | | | |
| | rectal bleeding or tearing during<br>or after a bowel movement | | | | | |
| | incomplete bowel movement,<br>like you didn't "finish" | | | | | |
| 1 | bowel movements that were too<br>hard | | | | | |
| | bowel movements that were too<br>small | | | | | |
| 11. | straining or squeezing to try to<br>pass bowel movements | | | | | |
| | feeling like you had to pass a<br>bowel movement but you<br>couldn't (false alarm) | | | | | |

Proprietary information of Janssen Research Foundation All rights reserved. 1997.